## Evaluation of EverLift in the Performance of Polypectomy for Polyps 4-9mm

NCT04551014

May 4, 2022

Shai Friedland, Principal Investigator Stanford University Stanford, California 94305

## Statistical analysis

In all analyses, P < 0.05 was considered significant. All tests were two-tailed. Student's t test was performed to evaluate the average of normally distributed continuous variables, and  $\chi^{[1]}$  test was performed to evaluate frequencies of categorical outcomes. Multivariate logistic regression was used to assess factors affecting complete resection of polyps, including use of EverLift<sup>TM</sup>, polyp size, Paris classification, time of polypectomy, attending performance of polypectomy, piecemeal resection, and polyp pathology. Analyses were performed using R Studio (RStudio, Inc.).

-

<sup>&</sup>lt;sup>1</sup> Repici et al (2018) Gastrointest Endosc 88(3):527-535.e5.